CLINICAL TRIAL: NCT00802672
Title: A Double-blind, Randomized, Parallel-group, Vehicle-controlled, Multi-center Study to Evaluate the Safety and Clinical Equivalence of a Generic Ciclopirox Olamine Cream to Ciclopirox Cream 0.77% in the Treatment of Tinea Pedis
Brief Title: Safety and Equivalence of a Generic Ciclopirox Olamine Cream Compared to the Reference Ciclopirox Cream 0.77% for the Treatment of Tinea Pedis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPL-302
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis; Ciclopirox Olamine
MeSH Terms: conditions — Tinea Pedis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Product (Experimental): Ciclopirox Olamine Cream 0.77%
  Interventions: Drug: Ciclopirox Olamine Cream
- Reference Product (Active Comparator): Loprox Cream 0.77%
  Interventions: Drug: Loprox Cream 0.77%
- Vehicle Product (Placebo Comparator): placebo of test product
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclopirox Olamine Cream — topical cream
  Arms: Test Product
Drug: Loprox Cream 0.77% — topical cream
  Other Names: Loprox Cream
  Arms: Reference Product
Drug: Placebo — topical cream
  Arms: Vehicle Product

SUMMARY:
The objectives of this study were to demonstrate comparable safety and efficacy of Ciclopirox Olamine Cream (Test Product) and Ciclopirox Cream 0.77% (Reference Product) in the treatment of subjects with tinea pedis, and to show the superiority of the active treatments over that of the vehicle.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 10 years of age, and otherwise healthy
* Clinically and mycologically confirmed diagnosis of symptomatic tinea pedis
* In good health with no clinically significant disease that might have interfered with study evaluations
* Study participant or legal guardian was willing and able to read and sign an IRB approved ICF, which included agreement to comply with all study requirements as indicated in the protocol. For subjects 10 to 17 years of age, an assent form for minors was completed.

Exclusion Criteria:

* History of hypersensitivity or allergy to ciclopirox
* Had any skin condition that would interfere with the diagnosis or assessment of tinea pedis
* Had a history of dermatophyte infecton unresponsive to antifungal treatment
* Had a history of alcoholism, drug abuse, or problems that would likely have made the subject unreliable for the study
* Had any condition or used any medication that, in the opinion of the Investigator, might have interfered with the conduct or results of the study or placed the prospective subject at increased risk
* Was unwilling to sign the informed consent
* Female who was pregnant or lactating

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2003-12; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Product: Ciclopirox cream
- Reference Product: Loprox Cream
- Vehicle Product: placebo
Period: Overall Study
Arm/Group | Test Product | Reference Product | Vehicle Product
Started | 224 | 226 | 111
Completed | 156 | 174 | 77
Not Completed | 68 | 52 | 34
Not completed — Lack of fungal pathogen at baseline | 56 | 43 | 25
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Protocol Violation | 2 | 1 | 1
Not completed — Lost to Follow-up | 5 | 5 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 2
Not completed — other | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Product | Reference Product | Vehicle Product | Total
Number analyzed (Participants) | 224 | 226 | 111 | 561
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 16 | 6 | 33
  Between 18 and 65 years | 194 | 189 | 92 | 475
  >=65 years | 19 | 21 | 13 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.2 (15.6) | 42.3 (15.6) | 43.1 (15.1) | 43.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 63 | 28 | 144
  Male | 171 | 163 | 83 | 417
Region of Enrollment [Number; unit: participants]
  United States | 224 | 226 | 111 | 561

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in Each Treatment Group With Therapeutic Success
Description: Both Mycological Cure (KOH wet mount negative and fungal culture negative) and Clinical Cure were required to achieve Therapeutic Success
Time Frame: 6 weeks
Population: Per protocol population
Measure: Number; unit: participants
Groups:
- Test Product: Ciclopirox Olamine Cream, USP
- Reference Product: Loprox® (ciclopirox) Cream 0.77%
- Vehicle Product: Vehicle
Arm/Group | Test Product | Reference Product | Vehicle Product
Number analyzed (Participants) | 141 | 166 | 68
participants | 70 | 95 | 3
Statistical Analysis 1: Comparison: Test Product vs Reference Product; Test type: Non-Inferiority or Equivalence — For the primary efficacy analysis, a 90% confidence interval was constructed for the difference in the Therapeutic Success rates between the Test Product and Reference Product at Visit 4/Week 6 (Follow-Up). The interval was calculated using Wald's method with Yates' continuity correction. Therapeutic equivalence (bioequivalence) was established if this 90% confidence interval was contained within the interval -0.20 to +0.20 (-0.20% to +0.20%); Wald's method with Yates' continuity; Mean Difference (Final Values) = 1, 90% CI 2-sided [-17.61 to 2.45]

2. Secondary Outcome: Proportion of Subjects With Mycological Cure
Description: Mycological Cure (KOH wet mount negative and fungal culture negative
Time Frame: 6 weeks
Population: per protocol population
Measure: Number; unit: participants
Arm/Group | Test Product | Reference Product | Vehicle Product
Number analyzed (Participants) | 141 | 166 | 68
participants | 107 | 133 | 9

3. Secondary Outcome: Proportion of Subjects With Clinical Cure
Description: Clinical Cure was defined as a signs and symptoms score of <1 for erythema; <1 for scaling; and 0 for pruritus, maceration, fissuring/cracking, and burning/stinging; as well as an assessment that no additional antifungal therapy was required to treat the subject's current episode of tinea pedis
Time Frame: 6 weeks
Population: per protocol population
Measure: Number; unit: participants
Arm/Group | Test Product | Reference Product | Vehicle Product
Number analyzed (Participants) | 141 | 166 | 68
participants | 82 | 106 | 9

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Test Product | Reference Product | Vehicle Product
Serious Adverse Events (participants affected / at risk) | 2/224 | 2/226 | 1/111
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product (N=224) | Reference Product (N=226) | Vehicle Product (N=111)
Pain secondary to head trauma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Near syncope (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other